CLINICAL TRIAL: NCT03938753
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2018_42
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sonova2018_42
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Hearing Loss; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phonak Audéo M90-T (Experimental): The Phonak Audéo M90-T is a Receiver-in-the-canal Hearing aid with direct connectivity functionality and a T-Coil from Phonak which will be fitted to the participants individual Hearing loss.
  Interventions: Device: Audéo M90-T

INTERVENTIONS:
Device: Audéo M90-T — Receiver in the canal (RIC) Hearing aid form Phonak which will be fitted to the participants individual Hearing loss.

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
In this study one CE-labeled Phonak Receiver-in-the-canal (RIC) devices is investigated. The experimental device will be investigated regarding Sound Quality perception ot the T-Coil program. A secondary objective of this study is the investigation of the Overall system stability in daily life situations. The experimental device contains direct connectivity functionality and a T-Coil. The combination of a wireless chip for Bluetooth streaming and a T-Coil in one housing can cause audible artifacts on the T-Coil, which shall be investigated within this study. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, moderate to severe Hearing loss)
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Willingness to wear Receiver in the canal hearing aids
* Informed Consent as documented by signature
* Owning a compatible smartphone

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Subjective perception of the T-Coil Sound Quality | 4 weeks
  The primary objective of this study is to measure that the overall sound Quality of the T-Coil program [subjective satisfaction rating on a scale from 0%-100% in 1% steps] of the investigational device is rated as at least as 60% or better [60% is the border between 'ok' and 'satisfied'] after a test period with daily life situations.

SECONDARY OUTCOMES:
Program switch-back workflow into T-Coil program | 4 weeks
  The number of incorrect switch-back occurences will be measured under laboratory conditions. A switch-back workflow is defined as the correct (re)activation of the T-Coil program, after an automatic program change into a streaming program. Due to an incoming phone call or due a start of audio streaming via Bluetooth, the investigational device will automatically switch into a streaming program. As soon as the Bluetooth stream stops, the investigation device must automatically toggle back into the T-Coil program (switch-back workflow).

OTHER OUTCOMES:
Observation of the system stability | 4 weeks
  Another objective of this study is the monitoring of the system stability during daily life situations. The investigational device will be worn for 4 weeks in home trial. Each investigational device will track the system stability in the background (unnoticeable for the HI-wearer). A log file of the system stability can be read out by the investigator. The system stability will be calculated by the amount of tracked system artefacts in relation to the overall wearing time. System artefacts are not or only hardly noticeable for the HI wearer, so that these system artefacts can only be tracked by reading out the data logging of the investigational device.
Sound Quality rating of T-Coil program under lab conditions | 4 weeks
  Another objective is the subjective perception of the Sound Quality of the T-Coil under laboratory condition. Subjects will rate the perceived Sound Quality of an audio file streamed via T-Coil on a scale from 'not at all' to 'excellent'.
Subjective perception of audio artefacts in T-Coil program | 4 weeks
  Another objective is to count the number of reports from subjects regarding audible artefacts in the T-Coil program after a home trial phase of 4 weeks. Audible artefacts are defined as any disturbing unnatural sounds which interfere with a streamed signal via T-Coil. Artefacts will be noted on a client questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland